CLINICAL TRIAL: NCT04425460
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase III Clinical Study Evaluating the Efficacy and Safety of Favipiravir in the Treatment of Adult Patients With COVID-19-Moderate Type
Brief Title: A Multi-center,Randomized,Double-blind,Placebo-controlled,Phase 3 Study Evaluating Favipiravir in Treatment of COVID19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS216C17(MRCT)
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, placebo-controlled (1:1) clinical study to explore the efficacy and safety of Favipiravir
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental): Favipiravir Tablets, 200 mg/tablet Favipiravir combined with supportive care recommended in the current National/Local guidelines. Favipiravir dosage and method of administration: Day 1: 1800mg, BID; Day 2 and thereafter: 600mg, TID, for a maximum of 14 days.
  Interventions: Drug: Favipiravir
- Placebo (Placebo Comparator): Placebo control group Favipiravir combined with supportive care recommended in the current National/Local guidelines
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Favipiravir — Favipiravir combined with supportive care recommended in the current National/Local guidelines. Favipiravir dosage and method of administration: Day 1 1800 mg x2; Day 2 up to a maximum of 14 days 600 mg x 3
  Arms: Favipiravir
Other: Placebo — Placebo combined with supportive care recommended in the current National/Local guidelines. Placebo dosage and method of administration: Day 1 1800 mg x2; Day 2 up to a maximum of 14 days 600 mg x 3
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, phase III clinical study to evaluate the efficacy of Favipiravir combined with supportive care for adult patients with COVID-19-Moderate type.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participating in the clinical study; fully understanding and being fully informed of the study and having signed the Informed Consent Form (ICF); willingness and capability to complete all the study procedures;
2. Age 18-75 years (inclusive) at the time of signing ICF;
3. Being confirmed with COVID-19-Moderate type according to Competent Authority and Ministry of Health and respective country guidelines and recommendations reported in Appendix 1 (a, b, c, d) to the present protocol. Based on comprehensive analysis and judgement taking into account both the epidemiological history and clinical manifestations, the diagnosis is to be confirmed for suspected cases or suspected cases/clinically diagnosed cases with all of the following etiological evidences:

   * Positivity in RT-PCR 2019-nCov test on respiratory tract specimens;
   * High homology with known gene sequence of 2019-nCov in viral gene sequencing on respiratory tract specimens.
4. Chest imaging (CT as first option or X-ray if CT not possible)-documented pneumonia; if CT cannot be performed, Pneumonia confirmed by X-ray may be used. The method of chest imaging pneumonia diagnosis must be consistent all through the study period;
5. Patients with pyrexia (axillary ≥37℃ or oral ≥ 37.5℃, or tympanic or rectal≥38℃) or either respiratory rate >24/min and <30/min or cough; For not hospitalized patients, the Investigator should maintain the detection method consistent through study period. In addition, the Investigator should maintain the data collection and quality compliant with GCP requirements.
6. The interval between symptoms onset and randomization is no more than 10 days; symptoms onset is primarily based on pyrexia, and can be based on cough or other related symptoms for patients without experiencing pyrexia following onset (it is strongly recommended that the interval between symptoms onset and randomization should not exceed 5 days);
7. For female subjects: evidence of post-menopause, or, for pre-menopause subjects, negative pre-treatment serum or urine pregnancy test. Menopause is defined as amenorrhea for at least 12 months without other medical cause, with the following age-specific requirements:

   * For female subjects aged <50 years: menopause for at least 12 months following withdrawal of exogenous hormonal therapy, with LH or FSH within the post-menopausal ranges, or having undergone any contraceptive surgery (bilateral oophorectomy or hysterectomy);
   * For female subjects aged ≥ 50 years: menopause for at least 12 months following withdrawal of exogenous hormonal therapy, or having undergone radiotherapy-induced oophorectomy with amenorrhea >1 year, or having undergone chemotherapy-induced menopause with amenorrhea>1 year, or having undergone any contraceptive surgery (bilateral oophorectomy or hysterectomy).
8. Eligible subjects of child-bearing age (male or female) must agree to take effective contraceptive measures (including hormonal contraception, barrier methods or abstinence) with his/her partner during the study period and for at least 3 months (in male) and 1 month (in female)following the last study treatment; in addition:

   1. For female participants of childbearing potential only highly effective methods (failure rate < 1 %) plus one barrier method is allowed throughout the period of relevant systemic exposure with Favipiravir. Double barrier methods alone are not considered as highly effective. Additionally, pregnancy testing at baseline only is not deemed sufficient and must be repeated more frequently, at least if clinical signs of pregnancy occur and at follow-up / end of study.
   2. male participants, if vasectomized or not, must wear a condom each time having heterosexual intercourse throughout the period of relevant systemic exposure with Favipiravir (as it is distributed to seminal fluid).
   3. male participant must be instructed not to have intercourse with pregnant women throughout the period of relevant systemic exposure with Favipiravir.
   4. For further details on contraception in clinical trials, please refer to the CTFG guidance: https://www.hma.eu/fileadmin/dateien/Human_Medicines/01- About_HMA/Working_Groups/CTFG/2014_09_HM A_CTFG_Contraception.pd
9. Not participating in any other drug clinical studies before completion of the present study.

Exclusion Criteria:

1. Where, in the opinion of the investigator, participation in this study will not be in the best interest of the subject, or any other circumstances that prevent the subject from participating in the study safely;
2. Refractory nausea, vomiting, or chronic gastrointestinal disorders, inability to swallow the study drug or having undergone extensive bowel resection which may affect adequate absorption of Favipiravir;
3. Severe liver disease: underlying liver cirrhosis or alanine aminotransferase (ALT)/aspartate aminotransferase (AST) elevated over 5 times the ULN;
4. Gout/history of gout or hyperuricemia (above the ULN);
5. Oxygen saturation (SPO2) ≤93% or arterial oxygen partial pressure (PaO2)/ fraction of inspired O2 (FiO2) ≤300 mmHg;
6. Known allergy or hypersensitivity to Favipiravir or any of its excipients, or to placebo excipients
7. Known severe renal impairment [creatinine clearance (CrCl) <30 mL/min] or having received continuous renal replacement therapy, hemodialysis or peritoneal dialysis;
8. Possibility of the subject being transferred to a non-study hospital within 72h;
9. Pregnant or lactating women;
10. Having used Favipiravir or participated in any other interventional drug clinical study within 30 days prior to first dose of study drug or having received treatments with other Investigational Medicinal Products (IMPs) or previous therapies within two weeks or five times the half-life of the drug, whichever is longer, must lead to exclusion
11. Persons, who were placed in an institution due to official or legal orders should be excluded
12. Persons, who are dependent on the sponsor, the investigator or the trial site, meaning that the voluntary nature of their consent is no longer guaranteed, must be excluded from participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to clinical recovery | 28 days
  The duration from start of treatment (Favipiravir or placebo) to normalization of pyrexia, respiratory rate and SPO2 and relief of cough (where there are relevant abnormal symptoms at enrolment) that is maintained for at least 72h.
  Criteria for normalization or relief:
  * Pyrexia (body temperature): axillary ≤37℃，or oral≤37.5℃，or rectal or tympanic
    ≤38℃;
  * Respiratory rate: ≤24/min without oxygen inhalation;
  * SPO2: >94% without oxygen inhalation;
  * Cough: Subject-perceived improvement or resolution of cough.

SECONDARY OUTCOMES:
Negativity in RT-PCR nucleic acid test | 28 days
  Time from randomization to negativity in RT-PCR nucleic acid test for 2019-nCov within 28 days of randomization;
Time from randomization to resolution of pyrexia | 28 days
  Time from randomization to resolution of pyrexia (defined the same as for the primary efficacy variable; applicable to subjects with pyrexia at enrolment) within 28 days of randomization;
Time from randomization to relief of cough | 28 days
  Time from randomization to relief of cough (defined the same as for the primary efficacy variable; applicable to subjects with cough at enrolment) within 28 days of randomization;
  It is recommended that the severity of cough be graded as per NCI-CTCAE v5.0:
  * Mild: Requires non-prescription treatment;
  * Moderate: Requires medication treatment; limits instrumental activities of daily living;
  * Severe: Limits self-care activities of daily living;
Incidence of deterioration/aggravation of pneumonia | 28 days
  Incidence of deterioration/aggravation of pneumonia (defined as SPO2≤93% or PaO2/FiO2 ≤300 mmHg or distressed RR≥30/min without oxygen inhalation and requiring oxygen therapy or more advanced breath support) within 28 days of randomization;
Time from randomization to relief of dyspnoea | 28 days
  Time from randomization to relief of dyspnoea (defined as subject-perceived improvement or resolution of dyspnoea; applicable to subjects with dyspnoea at enrolment) within 28 days of randomization;
Rate of auxiliary oxygen therapy or non-invasive ventilation | 28 days
  Rate of auxiliary oxygen therapy or non-invasive ventilation within 28 days of randomization;
ICU admission rate within 28 days of randomization | 28 days
  ICU admission rate within 28 days of randomization (except patients already enrolled in ICU which respect eligibility criteria);
All-cause mortality within 28 days of randomization. | 28 days
  All-cause mortality within 28 days of randomization.

CONTACTS AND LOCATIONS:
Locations (9):
- China (2):
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Shangcheng District
  - Peking University First Hospital, Beijing, Xicheng District
- Germany (2):
  - Department of Internal Medicine Pneumology and infectious diseases Neukölln Clinic, Berlin
  - Medical clinic and polyclinic IV Hospital of the University of Munich, München
- Romania (5):
  - Infectious Diseases Hospital Cluj-Napoca, Cluj-Napoca, Cluj
  - National Institute of Infectious Diseases "Prof.Dr.Matei Bals", Bucharest, Ilfov
  - "Dr.Victor Babes" Infectious Diseases and Pneumoftiziology Clinical Hospital Timisoara, Timișoara, Timiș County
  - Dr.Victor Babes Infectious Diseases and Pneumoftiziology Clinical Hospital Timisoara, Timișoara, Timiș County
  - Emergency County Hospital "Pius Brinzeu"Timisoara, Timișoara, Timiș County

IPD SHARING:
Plan to Share IPD: Undecided